CLINICAL TRIAL: NCT05914129
Title: Efficacy of Osteopathic Visceral Treatment on the Diaphragm, Stomach and Liver in Patients With Chronic Neck Pain
Brief Title: Efficacy of Osteopathic Visceral Treatment in Patients With Chronic Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OST1-008
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Cervical Pain
Keywords: Chronic Neck Pain; Diaphragm; Manual Therapy; Osteopathy; Visceral Techniques
MeSH Terms: conditions — Neck Pain | interventions — Contraceptive Devices, Female

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (GC) (Sham Comparator): To each volunteer, after 2 questionnaires, sham techniques will be performed to this group. The investigator will mimic the technique contacts without actually performing any type of tissue traction or compression, maintaining contact for the same amount of time described in the refered techniques. Following the technique, volunteers will answer the same 2 questionnaires shown previously.
  Interventions: Other: Sham technique
- Experimental Group A (GEA) (Experimental): To each volunteer, after 2 questionnaires, Diaphragm Stretching, Lower stomach mobilization and Liver pump techniques will be performed to this group. The diaphragm technique is performed 2 times with 1 minute interval, with the duration of 10 respiratory cycles. The lower stomach mobilization and liver pump techniques are performed one time, for 5 minutes each. Following the technique, volunteers will answer the same 2 questionnaires shown previously.
  Interventions: Other: Diaphragm, Stomach and Liver techniques
- Experimental Group B (GEB) (Experimental): To each volunteer, after 2 questionnaires, Lower stomach mobilization and Liver pump techniques will be performed to this group. These 2 techniques are the same ones as described for the experimental group A. Following the technique, volunteers will answer the same 2 questionnaires shown previously.
  Interventions: Other: Stomach and Liver techniques

INTERVENTIONS:
Other: Diaphragm, Stomach and Liver techniques — Diaphragm Stretching:
  The participant is seating down and the researcher will be behind, placing their hands on the inferior costal border. Cephalic traction is performed during inhalation, remaining during exhalation. Procedure is repeated 2 times, for 10 respiratory cycles, with 1-minute intervals.
  Inferior Mobilization of the Stomach:
  The participant is seating down with slight flexion of the torso, while the investigator stands behind them, placing the thumbs on the epigastric region. The volunteer will extend their body while the researcher performs a caudal traction. This procedure lasts 5 minutes.
  Liver Pump:
  Participant is laying on their back, and the investigator is standing on the participants side. The researcher places one hand on the right side inferior costal border posteriorly and the other one bellow the costal border anteriorly. Researcher compresses during exhalation and releases their hands abruptly during inhalation. This procedure lasts 5 minutes.
  Arms: Experimental Group A (GEA)
Other: Stomach and Liver techniques — In this group, techniques are the exact same as described previously but only liver and stomach ones will be performed.
  Arms: Experimental Group B (GEB)
Other: Sham technique — In the sham group, manual contact without any therapeutic intention will be performed in the same regions as the experimental groups. This contact will be maintained during the same amount of time as for the experimental group A.
  Arms: Control Group (GC)

SUMMARY:
This study aims to analyze the effects of visceral osteopathic treatment of the diaphragm, stomach and liver in the treatment of chronic neck pain.

DETAILED DESCRIPTION:
Cervical pain is a very common condition, whom can originate from bad posture, cervical tension, anxiety, depression and occupational or sportive activities. The influence of mobility and function changes of the abdominal viscera in the cervical region is a mechanism that is still poorly described in literature.

It is expected to find, through mechanical and neural pathways, that the visceral osteopathy treatment will have some effect on chronic neck pain.

This study intends to check the effects of the diaphragm stretching, inferior mobilization of the stomach and liver pump techniques (restoring mobility and normalizing function of the viscera) on the neck region, by employing some questionnaires/instruments.

During the present study, the effects of the visceral techniques will be analyzed in the following variables: Neck Disability Index (NDI), Numeric Pain Scale (NPS or END) and Global Pain Scale (GPS or EPGM).

ELIGIBILITY:
Inclusion Criteria:

* Pain in the posterior cervical region for more than 3 months;
* Knowing how to read and write;

Exclusion Criteria:

* Recent Cervicothoracic or Thoracoabdominal trauma (less than 6 months);
* Surgical procedure in the cervical region less than 6 months ago
* Surgical procedure in the abdominal region less than 6 months ago;
* Diagnosis of disc disease/radiculopathy;
* Rheumatic and/or neurological disease;
* Pregnancy status

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-08 (Estimated)

PRIMARY OUTCOMES:
Change in level of incapacity derived from neck pain 7 days after the intervention | 7 days after the intervention
  The Neck Disability Index questionnaire (NDI) will be the instrument used to evaluate the level of incapacity caused by neck pain. The questionnaire has 10 questions about the volunteers everyday life activities. There are 6 options to each question and the participant must choose the one that applies the most to their experience. The options selected will account for a score that goes from 0 to 50. The higher the number of the option, the more incapacity is felt and reported by the participant, meaning a worse outcome.
  This data will be collected by asking the volunteer their preferred option and writing it down.
Change in level of pain throughout the 7 days following the intervention | Once a day for the 7 days after the intervention
  The pain outcome will be measured according to the volunteers perception of pain in the cervical region by using the Numerical Pain Scale (NPS). This scale ranges from 0 to 10 and the participant must choose one number that best suits their level of current pain, 0 corresponding to "no pain" and 10 being "the worst pain imaginable to that participant". The higher the number, the worse the outcome.
  This data will be collected by asking the volunteer for the corresponding number and writing it down.

SECONDARY OUTCOMES:
Change in perception of the global conditions throughout the 7 days following the intervention | Once a day for the 7 days after the intervention
  One week after the intervention, the participants must answer the Global Perception of Change Scale (GPCS), which presents 7 options (from 1 to 7). The higher the number of the option, the more change was perceived and reported by the participant, meaning a better outcome. This instrument will guide the researcher to better understand if the intervention resulted in any kind of change to their initial condition.
  This data will be collected by asking the volunteer their preferred option and writing it down.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, Principal Investigator — Escola Superior de Saúde do Politécnico do Porto
Locations (1):
- Escola Superior da Saúde do Porto, Porto, Portugal

REFERENCES:
- [Background] Dal Farra F, Buffone F, Risio RG, Tarantino AG, Vismara L, Bergna A. Effectiveness of osteopathic interventions in patients with non-specific neck pain: A systematic review and meta-analysis. Complement Ther Clin Pract. 2022 Nov;49:101655. doi: 10.1016/j.ctcp.2022.101655. Epub 2022 Aug 11. PMID 35986986
- [Background] Franke H, Franke JD, Fryer G. Osteopathic manipulative treatment for nonspecific low back pain: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2014 Aug 30;15:286. doi: 10.1186/1471-2474-15-286. PMID 25175885
- [Background] Galaasen Bakken A, Eklund A, Hallman DM, Axen I. The effect of spinal manipulative therapy and home stretching exercises on heart rate variability in patients with persistent or recurrent neck pain: a randomized controlled trial. Chiropr Man Therap. 2021 Nov 29;29(1):48. doi: 10.1186/s12998-021-00406-0. PMID 34844625
- [Background] Gomez F, Escriba P, Oliva-Pascual-Vaca J, Mendez-Sanchez R, Puente-Gonzalez AS. Immediate and Short-Term Effects of Upper Cervical High-Velocity, Low-Amplitude Manipulation on Standing Postural Control and Cervical Mobility in Chronic Nonspecific Neck Pain: A Randomized Controlled Trial. J Clin Med. 2020 Aug 10;9(8):2580. doi: 10.3390/jcm9082580. PMID 32784959
- [Background] Groisman S, Malysz T, de Souza da Silva L, Rocha Ribeiro Sanches T, Camargo Bragante K, Locatelli F, Pontel Vigolo C, Vaccari S, Homercher Rosa Francisco C, Monteiro Steigleder S, Jotz GP. Osteopathic manipulative treatment combined with exercise improves pain and disability in individuals with non-specific chronic neck pain: A pragmatic randomized controlled trial. J Bodyw Mov Ther. 2020 Apr;24(2):189-195. doi: 10.1016/j.jbmt.2019.11.002. Epub 2019 Nov 13. PMID 32507144
- [Background] McCoss CA, Johnston R, Edwards DJ, Millward C. Preliminary evidence of Regional Interdependent Inhibition, using a 'Diaphragm Release' to specifically induce an immediate hypoalgesic effect in the cervical spine. J Bodyw Mov Ther. 2017 Apr;21(2):362-374. doi: 10.1016/j.jbmt.2016.08.015. Epub 2016 Sep 9. PMID 28532881
- [Background] Melo TM, Cunha FLL, Bezerra LMR, Salemi M, de Albuquerque VA, de Alencar GG, de Siqueira GR. Abdominal and Diaphragmatic Mobility in Adults With Chronic Gastritis: A Cross-Sectional Study. J Chiropr Med. 2023 Mar;22(1):11-19. doi: 10.1016/j.jcm.2022.05.004. Epub 2022 Jul 20. PMID 36844992
- [Background] Oliva-Pascual-Vaca A, Gonzalez-Gonzalez C, Oliva-Pascual-Vaca J, Pina-Pozo F, Ferragut-Garcias A, Fernandez-Dominguez JC, Heredia-Rizo AM. Visceral Origin: An Underestimated Source of Neck Pain. A Systematic Scoping Review. Diagnostics (Basel). 2019 Nov 12;9(4):186. doi: 10.3390/diagnostics9040186. PMID 31726685
- [Background] Rotter G, Fernholz I, Binting S, Keller T, Roll S, Kass B, Reinhold T, Willich SN, Schmidt A, Brinkhaus B. The effect of osteopathic medicine on pain in musicians with nonspecific chronic neck pain: a randomized controlled trial. Ther Adv Musculoskelet Dis. 2020 Dec 10;12:1759720X20979853. doi: 10.1177/1759720X20979853. eCollection 2020. PMID 33354233
- [Background] Silva ACO, Biasotto-Gonzalez DA, Oliveira FHM, Andrade AO, Gomes CAFP, Lanza FC, Amorim CF, Politti F. Effect of Osteopathic Visceral Manipulation on Pain, Cervical Range of Motion, and Upper Trapezius Muscle Activity in Patients with Chronic Nonspecific Neck Pain and Functional Dyspepsia: A Randomized, Double-Blind, Placebo-Controlled Pilot Study. Evid Based Complement Alternat Med. 2018 Nov 11;2018:4929271. doi: 10.1155/2018/4929271. eCollection 2018. PMID 30534176
- [Background] Silva ACO, Oliveira CS, Biasotto-Gonzalez DA, Fumagalli MA, Politti F. Visceral Manipulation Decreases Pain, Increases Cervical Mobility and Electromyographic Activity of the Upper Trapezius Muscle in Non-Specific Neck Pain Subjects with Functional Dyspepsia: Two Case Reports. Int J Ther Massage Bodywork. 2019 Jun 1;12(2):25-30. eCollection 2019 Jun. PMID 31191786